CLINICAL TRIAL: NCT02943304
Title: Risk Evaluation of Fetal Nervous System and Neurodevelopment Disorders in Infants of Women Exposed to Zika Virus Infection During Pregnancy
Brief Title: Neurodevelopment Outcome of Newborns Exposed to Zika Virus (ZIKV) in Utero
Acronym: ZENI
Status: Completed | Type: Observational
Sponsor: Universidad Industrial de Santander (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Mario Augusto Rojas, Professor of Pediatrics, Universidad Industrial de Santander
Other Study IDs: 4110
Record Dates: First submitted 2016-10-20; First posted 2016-10-24 (Estimated); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Microcephaly; Mental Retardation
Keywords: Pregnancy; Fetal Development; Child Development; Developmental Disabilities; Zika Virus Infection
MeSH Terms: conditions — Microcephaly; Intellectual Disability; Developmental Disabilities; Zika Virus Infection | interventions — Urination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Maternal serum Amniotic Fluid Urine CSF
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Exposed: Symptomatic pregnant women with positive RT-PCR ZIKV in serum or urine, or a positive serologic test specific for ZIKV
  Interventions: Other: Symptomatic pregnant women with positive RT-PCR ZIKV in serum or urine, or a positive serologic test specific for ZIKV
- Unexposed: Asymptomatic pregnant women with a negative RT-PCR ZIKV in serum and urine, and a negative specific serology for ZIKV at enrollment into the study and at the time of delivery

INTERVENTIONS:
Other: Symptomatic pregnant women with positive RT-PCR ZIKV in serum or urine, or a positive serologic test specific for ZIKV
  Groups: Exposed

SUMMARY:
This prospective cohort study will determine the natural history of fetal exposure to Zika virus (ZIKV) and its effects on the fetus and newborn with emphasis on neurodevelopment outcome. Exposure of the fetus will be determined by maternal symptomatology, RT-PCR ZIKV (blood and urine) and serologic test specific for ZIKV. Neonates will be classified according to trimester of infection and as exposed and unexposed to ZIKV.

DETAILED DESCRIPTION:
Infection with Zika Virus (ZIKV) is an emerging disease in South America and a serious public health problem due to a high prevalence of one of the vectors that transmit the virus, Aedes Aegypti, and the severe and sometimes fatal complications that can be generated in the fetus of women infected by the virus during their pregnancy. Retrospective studies have shown an association with microcephaly, cerebral calcifications, dysgenesis of the corpus callosum, and other anomalies of the central nervous system (CNS). The high risk of neurodevelopmental impairment in the exposed newborn is a major concern.

The epidemiologic and neurobiological evidence supporting the link between infection of pregnant women, trimester of infection, and the development of such anomalies in the fetus is growing to the extent that the Center for Disease Control has officially made a statement supporting this association. Although the dimension of the public health impact is still unknown, limited prospective data makes counseling of pregnant women difficult, especially when they are considering termination of pregnancy.

Given that evidence supporting the neurotropic quality of ZIKV and the potential variations of the effect the virus may have on the developing fetal brain according to the gestational age of infection, we have designed a prospective cohort study to determine whether exposure of the fetus to ZIKV in symptomatic mothers results in fetal CNS anomalies and/or impaired neurodevelopmental outcome of the newborn. As a secondary aim we will determine the effect gestational age has on severity of CNS anomalies and neurodevelopmental outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women who on their first prenatal visit (independent of gestational age) confirm through a pre-designed questionnaire that they have had any symptom(s) compatible with ZIKV infection (rash [exanthema or sprout], conjunctivitis, arthralgia or myalgia, fever). Pregnant women with an affirmative response will be categorized in two groups:

   * Acute Infection: symptoms of ZIKV infection that occurred within the previous 14 days of the day the pregnant women attended her prenatal visit.
   * Late Infection: symptoms of ZIKV infection that occurred more then 14 days from her prenatal visit. Gestational age of onset of symptomatology will be documented at this time.
2. Pregnant women without symptoms of ZIKV infection who have a negative RT-PCR for ZIKV and a negative specific serologic test for ZIKV at initial prenatal visit with normal prenatal evaluation. These pregnant women will be selected from non high-risk delivery services.

Exclusion Criteria:

1. Eligible pregnant women that refuse to sign consent for participation in the ZEN Initiative.
2. Enrolled pregnant women that withdraw their consent to participate at any time in the study.

Ages: 13 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: ZIKV symptomatic and asymptomatic pregnant women in hyper endemic areas of ZIKV in Colombia
Sampling Method: Non-Probability Sample
Enrollment: 284 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Neurodevelopmental Outcome | 24 months corrected age
  Bayley Scales of Infant and Toddler Development Third Edition

SECONDARY OUTCOMES:
Fetal CNS Impairment | Until Birth
  Prenatal Level III Ultrasound Identification of Fetal CNS Abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Mario A Rojas, MD, MPH, Principal Investigator — Professor of Pediatrics; Luz A Gutierrez, MD, Study Director — Universidad Industrial de Santander; Luis A Diaz, MD, MSc, Study Chair — Universidad Industrial de Santander
Locations (1):
- Hospital Universitario de Santander, Bucaramanga, Santander Department, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diaz-Martinez LA, Rojas MA, Pinilla-Garcia LS, Becerra-Mojica CH, Perez-Vera LA, Gutierrez-Sanchez LA, Contreras-Garcia GA, Rueda-Ordonez CG, Villar L. Neurodevelopmental outcome of infants without central nervous system anomalies born to symptomatic RT-PCR ZIKV positive women. PLoS Negl Trop Dis. 2022 Mar 7;16(3):e0009854. doi: 10.1371/journal.pntd.0009854. eCollection 2022 Mar. PMID 35255097